CLINICAL TRIAL: NCT00823251
Title: IlluminOss Medical- Photodynamic Bone Stabilization System- International Study
Brief Title: IlluminOss Hand Fracture International Clinical Feasibility Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlluminOss Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILLUM-OUS-2008-001
Record Dates: First submitted 2008-12-30; First posted 2009-01-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Orthopedic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IlluminOss device (Experimental): IlluminOss bone-pin device
  Interventions: Device: IlluminOss device

INTERVENTIONS:
Device: IlluminOss device — The IlluminOss™ Bone Stabilization System is designed to deliver the device to the fracture site via the medullary canal of the bone using percutaneous techniques. Once the device is in place and has spanned the fracture site, the device is expanded and hardened to reduce and stabilize the fracture, to aid in the support and healing of the bone fracture by primary callous formation and remodeling.

SUMMARY:
The purpose of this study is to assess the initial safety and technical feasibility of the IlluminOss System in the treatment of fractures of bones in the hand.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Patient or his/her legal guardian understands the nature of the procedure and is willing to comply with associated follow-up evaluations, and provides written informed consent prior to the procedure
* Female patients must be of non-child bearing potential, or have a negative pregnancy test within prior 48 hours
* Acute fracture of metacarpal or phalangeal bone(s) that requires reduction and internal fixation
* Fracture has occurred within past 3 weeks
* Fracture types: transverse, short oblique, or any fracture pattern in which the comminuted segment is equal to or less than the diameter of the bone at fracture site

Exclusion Criteria:

* Patient is pregnant, lactating or female patients who intend to become pregnant during the course of the study
* Patient has experienced a crush, mangling, or burn type injury
* Patient has probable history of infection or confirmed infection at baseline
* Patient has previous diagnosis of a significant bone disorder that may impair bone healing
* Patient has a life expectancy of < 26 weeks
* Pathological fracture secondary to tumor
* Open fracture of Gustilo-Anderson Type II or III

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Technical Success: Successful implantation of an IlluminOss bone-pin via percutaneous techniques at the target fracture location. | Immediately post-surgery

SECONDARY OUTCOMES:
Rate of Fracture Union | 180 day
Rate of Anatomic Alignment | 180 Day
Functionality Score | 180 Day
Grip Strength | 180 Day
Range of Motion | 180 day
Incidence of Reintervention of Target Fracture | 180 Day
Bone Pin Migration | 180 Day
Adverse Event Rate | 180 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Trabajador, Santiago, Chile